CLINICAL TRIAL: NCT05151315
Title: Component Migration, Polyethylene Wear, and Joint Inflammation of the Evolution Versus Evolution NitrX Total Knee Arthroplasty System
Brief Title: NitrX Total Knee Arthroplasty RSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Principal Investigator, Edward Vasarhelyi, Orthopaedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 119937
Record Dates: First submitted 2021-11-05; First posted 2021-12-09 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Total Knee Arthroplasty; Knee Osteoarthritis; Radiostereometric Analysis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolution Total Knee Arthroplasty system (Active Comparator): Patients will undergo total knee arthroplasty with the Evolution Total Knee System
  Interventions: Device: Total Knee Arthroplasty with Evolution Knee System
- Evolution with NitrX Total Knee Arthroplasty system (Experimental): Patients will undergo total knee arthroplasty with the NitrX Evolution Total Knee System which has the specialized protective coating
  Interventions: Device: Total Knee Arthroplasty with Evolution® NitrX™ Knee System

INTERVENTIONS:
Device: Total Knee Arthroplasty with Evolution® NitrX™ Knee System — Patients will receive cemented Evolution knee system with NitrX coating for their total knee arthroplasty.
  Arms: Evolution with NitrX Total Knee Arthroplasty system
Device: Total Knee Arthroplasty with Evolution Knee System — Patients will receive cemented Evolution knee system without NitrX coating for their total knee arthroplasty.
  Arms: Evolution Total Knee Arthroplasty system

SUMMARY:
Metal hypersensitivity is a recognized complication in some patients following total joint arthroplasty. This can result in a reaction to metal particles from the implants placed in the joint and cause tissue injury. The Evolution® NitrX™ (MicroPort Orthopaedics, Memphis, TN) knee implant was designed with the addition of a coating meant to create a barrier against the release of metal ions. The primary purpose of this study is to compare the Evolution and Evolution NitrX implant (implants your surgeon uses in total knee arthroplasty surgery). This study will compare the stability of these knee implants (any movement the implant makes after surgery) through the use of specialized xrays, called "radiostereometric analysis" (RSA for short). The investigators will also compare levels of circulating metal particles with blood draws and the effects of any circulating metal with MR imaging. The investigators will also be looking at the participants clinical outcomes using joint function and patient satisfaction questionnaires. A total of 50 patients will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee indicating primary total knee arthroplasty
* Varus knee deformity of 0 to 10 degrees
* Sufficient ligamentous function to warrant retention of the posterior cruciate ligament
* Between ages of 21 and 80 inclusive
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent
* No contraindications to Magnetic Resonance Imaging (MRI)

Exclusion Criteria:

* Active or previous infection
* Medical condition precluding major surgery
* Inflammatory arthropathy
* Prior Patellectomy
* PCL deficiency
* Major Coronal plane deformity
* Valgus deformity
* Bone defects requiring augments, cones and/or stemmed implants

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Implant Migration (Tibial Component) | 2 years
  Model based Radiostereometric Analysis (RSA, specialized Xrays) will be used to register the location of the tibial implant components during supine and standing exams and measure implant movement. Changes throughout the different time points of potential tibial migration, with the use of the tibial bone beads, will be measured in millimeters.

SECONDARY OUTCOMES:
Implant Migration (Femoral Component) | 2 years
  Model based Radiostereometric Analysis (specialized Xrays) will be used to register the location of the femoral components during supine and standing exams and measure implant movement. Changes throughout the different time points of potential femoral migration, with the use of the femoral bone beads, will be measured in millimeters.

OTHER OUTCOMES:
Wear Rates | 2 weeks (baseline), 6 weeks, 3 months, 6 months, 1 year, and 2 years.
  Model based Radiostereometric Analysis (specialized Xrays) will be used to register the location of the femoral and tibial components in both standing and supine exams where the minimum joint space width between components on the medial and lateral condyles can be calculated as a measurement (in millimeters) of polyethylene wear.
Circulating metal levels | Pre-operative, 1 and 2 years post-operatively.
  Patients will have blood drawn and the levels of circulating cobalt, chromium, and nickel will be measured in whole blood. One vial of blood will be drawn from the patient (in milliliters).
Synovial Joint Inflammation observation | 2 Years
  Patients will complete an MRI exam using metal artefact reduction sequences. Scans will be evaluated and scored for synovial inflammation and fibrosis, indicative of reactions to metal debris, and the presence of fibrous tissue at the bone-cement-implant interface, indicative of component loosening.
Knee Injury and Osteoarthritis Outcome score (KOOS) | Pre-operative, 3 months, 1 year, and 2 year post-operative
  Patient reported outcome measure. Holds 42 items that asks patient about pain, functional daily living, and sport and recreation. Questionnaire measures levels in frequency (never to always) and severity (none to extreme). Scores are from 0-100, with higher scores indicating no knee problems.
Forgotten Joint Score (FJS) | Pre-operative, 3 months, 1 year, and 2 year post-operative
  Patient reported outcome measure observing the ability of a patient to forget about a joint due to successful treatment. Contains 12 items with frequency level measurement (never to mostly). The higher the score (0-100), the less aware the patient is of their affected joint when performing daily activity.
Veterans-Rand 12 Item Health Survey (VR-12) | Pre-operative, 3 months, 1 year, and 2 year post-operative
  Patient reported outcome measure observing physical and mental health status of patient. Contains 14 items measuring levels of severity (excellent to poor) and frequency (None of the time to Yes, all of the time). Higher scores indicate higher quality of life and vice versa.
European Quality of Life - 5 Dimension (EQ-5D) | Pre-operative, 3 months, 1 year, and 2 year
  Patient reported outcome measure. Standardized 5 item instrument measuring generic health status of patient. The EQ5D uses a Likert scale which assesses five states (mobility, self care, usual care, pain and discomfort and anxiety and depression) at five different levels - none(0), slight(1), moderate(2), severe(3) or unable to perform(5). Levels are coded 1-5 and an index score is then generated. Higher scores indicate higher health status of patient.
Metal Exposure/Sensitivity | Pre-operative
  Patient reported outcome measure. Screening tool for noting pre-operative environmental metal exposures. Questionnaire contains Yes or No questions. Higher scores would indicate greater exposure and/or metal sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Edward M Vasarhelyi, MD, Principal Investigator — London Health Sciences Centre; Matthew Teeter, PhD, Principal Investigator — London Health Science Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pijls BG, Plevier JWM, Nelissen RGHH. RSA migration of total knee replacements. Acta Orthop. 2018 Jun;89(3):320-328. doi: 10.1080/17453674.2018.1443635. Epub 2018 Mar 6. PMID 29508661
- [Background] Teeter MG, Marsh JD, Howard JL, Yuan X, Vasarhelyi EM, McCalden RW, Naudie DDR. A randomized controlled trial investigating the value of patient-specific instrumentation for total knee arthroplasty in the Canadian healthcare system. Bone Joint J. 2019 May;101-B(5):565-572. doi: 10.1302/0301-620X.101B5.BJJ-2018-1323.R1. PMID 31038991
- [Background] Teeter MG, Thoren J, Yuan X, McCalden RW, MacDonald SJ, Lanting BA, Naudie DD. Migration of a cemented fixed-bearing, polished titanium tibial baseplate (Genesis II) at ten years : a radiostereometric analysis. Bone Joint J. 2016 May;98-B(5):616-21. doi: 10.1302/0301-620X.98B5.36865. PMID 27143731
- [Background] Teeter MG, Perry K, Yuan X, Howard JL, Lanting BA. The Effects of Resection Technique on Implant Migration in Single Radius Posterior-Stabilized Total Knee Replacement. J Knee Surg. 2020 Jan;33(1):78-83. doi: 10.1055/s-0038-1676462. Epub 2018 Dec 18. PMID 30562833
- [Background] Sealed Envelope Ltd.2012.Power calculator for continuous outcome non0-inferiority trial.[Online] Available from: https://www.sealedenvelope.com/power/continuous-noninferios/[Accessed Thu Jan 14 2021].
- [Background] van Ijsseldijk EA, Valstar ER, Stoel BC, de Ridder R, Nelissen RG, Kaptein BL. Measuring polyethylene wear in total knee arthroplasty by RSA: differences between weight-bearing and non-weight-bearing positioning. J Orthop Res. 2014 Apr;32(4):613-7. doi: 10.1002/jor.22579. Epub 2014 Jan 7. PMID 24395396
- [Background] Teeter MG, Wihlidal J, McCalden RW, Yuan X, MacDonald SJ, Lanting BA, Naudie DD. Radiostereometric Analysis Permits In Vivo Measurement of Very Small Levels of Wear in TKA. Clin Orthop Relat Res. 2019 Jan;477(1):80-90. doi: 10.1097/CORR.0000000000000399. PMID 30794231
- [Background] Gascoyne T, Parashin S, Teeter M, Bohm E, Laende E, Dunbar M, Turgeon T. In vivo wear measurement in a modern total knee arthroplasty with model-based radiostereometric analysis. Bone Joint J. 2019 Nov;101-B(11):1348-1355. doi: 10.1302/0301-620X.101B11.BJJ-2018-1447.R2. PMID 31674253
- [Background] Koff MF, Burge AJ, Potter HG. Clinical magnetic resonance imaging of arthroplasty at 1.5 T. J Orthop Res. 2020 Jul;38(7):1455-1464. doi: 10.1002/jor.24606. Epub 2020 Feb 4. PMID 31975444
- [Background] Attard V, Li CY, Self A, Mann DA, Borthwick LA, O'Connor P, Deehan DJ, Kalson NS. Quantification of intra-articular fibrosis in patients with stiff knee arthroplasties using metal-reduction MRI. Bone Joint J. 2020 Oct;102-B(10):1331-1340. doi: 10.1302/0301-620X.102B10.BJJ-2020-0841.R1. PMID 32993344
- [Background] Heyse TJ, Chong le R, Davis J, Boettner F, Haas SB, Potter HG. MRI analysis of the component-bone interface after TKA. Knee. 2012 Aug;19(4):290-4. doi: 10.1016/j.knee.2011.05.011. Epub 2011 Jul 8. PMID 21741843